CLINICAL TRIAL: NCT04703725
Title: The Effect of the Counseling on Women in In Vitro Fertilization (IVF) Process on Emotional Capacity and Well-Being
Brief Title: The Effect of IVF Counseling on Psychosocial Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ergul Aslan, Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9199
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Infertility; Psychological Distress; Infertility, Female; Depression, Anxiety; Nurse's Role
MeSH Terms: conditions — Infertility; Infertility, Female; Depression; Anxiety Disorders | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Experimental Design
Who Masked: Participant
Masking Description: In the single-blind method, subjects do not know which of the experimental or control groups they were selected and therefore which method was applied to them.The researcher knows the subjects selected for the experimental and control groups, and therefore which method was applied to which subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Infertile women recruited to the experimental group by randomization will be given a counseling program including psychosocial care in addition to routine (drug explanation during the treatment, preparation before the egg pick up and embryo transfer and post operative care). IVF treatment
  Interventions: Behavioral: Psychosocial Care
- Control Group (No Intervention): Routine (drug explanation during the treatment, preparation before the egg pick up and embryo transfer and post operative care) IVF treatment will be applied to infertile women who are randomized to the control group.

INTERVENTIONS:
Behavioral: Psychosocial Care — 1. First Follow-Up: One of the implementation of the module
  2. Second Follow-up: Implementation of the second module; Breathing Exercises and EFT
  3. Third Follow-up: Emotional preparation about egg pick up process, individual application of coping methods
  4. Fourth Follow-up: Implementation of the second module; Briefing about Breathing Exercises and EFT embryo transfer process
  5. Fifth Follow-up: Implementation of the second module; Breathing Exercises and EFT
  6. Sixth Follow-up: Individual application of coping methods until the learning process of pregnancy test result
  7. Seventh Follow-up: Providing information about the first periods of pregnancy after treatment resulting in pregnancy and providing information about the psychosocial problems that may be encountered. Identifying psychosocial problems that may be encountered after unsuccessful treatment and individual application of coping methods to help cope.
  Other Names: First Follow-Up; Second Follow-up; Third Follow-up; Fourth Follow-up; Fifth Follow-up; Sixth Follow-up; Seventh Follow-up
  Arms: Experimental Group

SUMMARY:
In this study, İt was aimed to determination of the effect of counseling given in accordance with the Roy Adaptation Model in women in the in vitro fertilization (IVF) process on emotional capacity and well-being.

DETAILED DESCRIPTION:
The study will be conducted in the Infertility clinic of a medical school hospital. The study included women receiving IVF treatment. In the pre-initial evaluation, "Introductory Information Form, Screening on distress in fertility treatment (SCREENIVF), Infertility Stress, Life Quality Scale for Persons with Fertility Problems(FertiQol), Subjective Units of Distress Scale-SUD application is planned. A "Consultancy Program" will be applied to the experimental group in the form of two modules in addition to drug applications, egg pick up and embryo transfer before, during and after clinical routine health care. The first module of the counseling program is the definition of infertility, the treatment process, its effects on the life process and coping methods. The second module includes the application of breath awareness and Emotional Freedom Technique (EFT) within the scope of coping methods with infertility stress. Emotional Freedom Technique-EFT is an energy psychotherapy based on the principle that each limiting thought, disturbing emotion and memory of an individual disrupts the energy flow in the body and creates congestion. This technique, the stimulation on the meridian system by focusing on the thought, disturbing emotion or memory that prevents the individual (often by touching) regulates the energy flow and provides the individual to relax. With breath awareness, beneficial results can be obtained, such as physical, sensory and mental control, life-facilitating techniques, individual and social awareness, re-existence and raising the level of consciousness. Within the scope of the counseling program, a total of seven follow-ups will be made, five-to-one, via two phone calls. On the day of follicle development (2nd Follow-up), Egg Pick up Procedure (4th Follow-up) and Embryo transfer (5th Follow-up), the patient will be given breathing exercises and EFT and Subjective Units of Distress Scale will be scored. The control group will continue clinical routine health care and will be followed up on the first day of IVF treatment (1st follow-up) and on the seventh day of embryo transfer (2nd follow-up). For ethical reasons, a consultancy program will be applied to the control group after the second follow-up. Data collection tools will be applied again to both groups in the final evaluation.

ELIGIBILITY:
Inclusion Criteria:

* IVF treatmant
* Women
* Women aged18-40 years
* Sign the informed consent form

Exclusion Criteria:

* Having a psychiatric diagnosis /
* Having a situation that prevents communication (language, etc.)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women who are infertile and receiving if treatment
Enrollment: 85 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Screening on distress in fertility treatment | Measurement for each group in the beginning of the IVF treatment
  Anxiety (state anxiety, trait anxiety), Depression, Social support, Cognitions regarding fertility problems are measured using screening on distress in fertility treatment (SCREENIVF).
Screening on distress in fertility treatment | Measurement for each group seven days after embryo transfer
  Anxiety (state anxiety, trait anxiety), Depression, Social support, Cognitions regarding fertility problems are measured using screening on distress in fertility treatment (SCREENIVF).
Infertility Stress | Measurement for each group in the beginning of the IVF treatment
  Personal stress, marital stress, and social stress are measured using The Fertility Problem Stress Inventory
Infertility Stress | Measurement for each group seven days after embryo transfer
  Personal stress, marital stress, and social stress are measured using The Fertility Problem Stress Inventory
Life Quality Scale for Persons with Fertility Problems | Measurement for each group in the beginning of the IVF treatment
  Life Quality Scale for Persons with Fertility Problems (FertiQol) is used to measure the effect of quality and accessibility of treatment on quality of life.
Life Quality Scale for Persons with Fertility Problems | Measurement for each group seven days after embryo transfer
  Life Quality Scale for Persons with Fertility Problems (FertiQol) is used to measure the effect of quality and accessibility of treatment on quality of life.
Subjective Units of Distress Scale | The day follicle development is followed
  Applied to the experimental group. Before starting the application in energy therapies, the problem is evaluated with the severity of the discomfort. It is the subjective evaluation of the discomfort felt by the individual.
Subjective Units of Distress Scale | Egg pick up procedure day
  Applied to the experimental group.Before starting the application in energy therapies, the problem is evaluated with the severity of the discomfort. It is the subjective evaluation of the discomfort felt by the individual.
Subjective Units of Distress Scale | Embryo transfer day
  Applied to the experimental group.Before starting the application in energy therapies, the problem is evaluated with the severity of the discomfort. It is the subjective evaluation of the discomfort felt by the individual.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University-Cerrrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research article will be shared after publication

REFERENCES:
- [Background] Van den Broeck U, Emery M, Wischmann T, Thorn P. Counselling in infertility: individual, couple and group interventions. Patient Educ Couns. 2010 Dec;81(3):422-8. doi: 10.1016/j.pec.2010.10.009. Epub 2010 Nov 13. PMID 21075589
- [Background] Gameiro S, Boivin J, Dancet E, de Klerk C, Emery M, Lewis-Jones C, Thorn P, Van den Broeck U, Venetis C, Verhaak CM, Wischmann T, Vermeulen N. ESHRE guideline: routine psychosocial care in infertility and medically assisted reproduction-a guide for fertility staff. Hum Reprod. 2015 Nov;30(11):2476-85. doi: 10.1093/humrep/dev177. Epub 2015 Sep 7. PMID 26345684
- [Background] Ockhuijsen HDL, van Smeden M, van den Hoogen A, Boivin J. Validation study of the SCREENIVF: an instrument to screen women or men on risk for emotional maladjustment before the start of a fertility treatment. Fertil Steril. 2017 Jun;107(6):1370-1379.e5. doi: 10.1016/j.fertnstert.2017.04.008. Epub 2017 May 10. PMID 28501369
- [Background] Homan GF, Davies M, Norman R. The impact of lifestyle factors on reproductive performance in the general population and those undergoing infertility treatment: a review. Hum Reprod Update. 2007 May-Jun;13(3):209-23. doi: 10.1093/humupd/dml056. Epub 2007 Jan 5. PMID 17208948
- [Background] Verhaak CM, Smeenk JM, van Minnen A, Kremer JA, Kraaimaat FW. A longitudinal, prospective study on emotional adjustment before, during and after consecutive fertility treatment cycles. Hum Reprod. 2005 Aug;20(8):2253-60. doi: 10.1093/humrep/dei015. Epub 2005 Apr 7. PMID 15817584
- [Background] Frederiksen Y, Farver-Vestergaard I, Skovgard NG, Ingerslev HJ, Zachariae R. Efficacy of psychosocial interventions for psychological and pregnancy outcomes in infertile women and men: a systematic review and meta-analysis. BMJ Open. 2015 Jan 28;5(1):e006592. doi: 10.1136/bmjopen-2014-006592. PMID 25631310